CLINICAL TRIAL: NCT01401244
Title: A Trial to Examine the Bioequivalence of Norditropin® Versus Genotropin® in Healthy Adult Volunteers
Brief Title: Bioequivalence of Two Somatropin Products (Norditropin® Versus Genotropin®) in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GH-3939; U1111-1121-3640 (Other: WHO)
Record Dates: First submitted 2011-07-20; First posted 2011-07-25 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Genetic Disorder; Prader-Willi Syndrome; Growth Disorder; Idiopathic Short Stature; Healthy
MeSH Terms: conditions — Genetic Diseases, Inborn; Prader-Willi Syndrome; Growth Disorders | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Norditropin® (Experimental)
  Interventions: Drug: somatropin
- Genotropin® (Active Comparator)
  Interventions: Drug: somatropin

INTERVENTIONS:
Drug: somatropin — A single dose 4.0 mg administered subcutaneously (under the skin) via Norditropin® FlexPro® pen
  Arms: Norditropin®
Drug: somatropin — A single dose 4.0 mg administered subcutaneously (under the skin) via Genotropin® Pen 12
  Arms: Genotropin®

SUMMARY:
This trial is conducted in United States of America (USA). The aim of this trial is to examine the bioequivalence of Norditropin® versus Genotropin® in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18.0-27.0 kg/m^2 (both inclusive)
* Considered generally healthy upon completion of medical history, physical examination, vital signs, screening laboratory results, and electrocardiogram (ECG), as judged by the Investigator (trial physician)

Exclusion Criteria:

* The receipt of any investigational medicinal product within 1 month prior to this trial
* Current or previous treatment with growth hormone or IGF-I (insulin-like growth factor-I)
* Female of childbearing potential who is pregnant, breast-feeding or intends to become pregnant or is not using adequate contraceptive methods (adequate contraceptive measures as required by local law or practice) for the duration of the trial
* Known presence or history of malignancy
* Diabetes mellitus
* Use of pharmacologic doses of glucocorticoids
* Use of anabolic steroids
* History of drug or alcohol abuse

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2011-07-14 (Actual); Primary Completion 2011-09-27 (Actual); Study Completion 2011-09-27 (Actual)

PRIMARY OUTCOMES:
Area under the serum hGH (human growth hormone) concentration-time curve | from 0 to the time of the last quantifiable concentration over a 24-hour sampling period
Maximum observed serum hGH concentration | over a 24-hour sampling period

SECONDARY OUTCOMES:
Area under the effect (IGF-I) curve | from time 0 to the time of the last concentration (AUEC0-t) over a 96-hour sampling period
Maximum IGF-I effect (Emax) | over a 96-hour sampling period
The frequency of adverse events (AE) | from screening (3-14 days before first dose of trial product) to follow-up period (day 17 after first dose of trial product)
The frequency of injection site reaction | from the time of injection of the trial product (day 1 and 13, respectively) to follow-up during the two dosing periods (day 5 and 17, respectively)
Abnormal hematology laboratory parameters | from screening (3-14 days before first dose of trial product) to follow-up period (day 17 after first dose of trial product)
Abnormal biochemistry laboratory parameters | from screening (3-14 days before first dose of trial product) to follow-up period (day 17 after first dose of trial product)
Abnormal findings in physical examinations | from screening (3-14 days before first dose of trial product) to follow-up period (day 17 after first dose of trial product)
Vital signs | from screening (3-14 days before first dose of trial product) to follow-up period (day 17 after first dose of trial product)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Evansville, Indiana, United States

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com